CLINICAL TRIAL: NCT02080351
Title: A Simple Cognitive Task to Reduce the Build-Up of Flashbacks After a Road Traffic Accident: A Randomised Controlled Study in an Emergency Department
Brief Title: A Simple Cognitive Task to Reduce the Build-Up of Flashbacks After a Road Traffic Accident
Acronym: SCARTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other); National Institute for Health Research, United Kingdom (Other Government); Medical Research Council Cognition and Brain Sciences Unit (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12/SC/0485
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Post-traumatic Stress Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simple cognitive task (Experimental): A memory reactivation cue followed by playing the computer game "Tetris"
  Interventions: Behavioral: Simple cognitive task
- Usual care (No Intervention): Usual care in the emergency department

INTERVENTIONS:
Behavioral: Simple cognitive task
  Arms: Simple cognitive task

SUMMARY:
This research study is designed to investigate the effects of a simple cognitive task (a memory reactivation cue following by playing the computer game "Tetris") on flashbacks and other post-traumatic stress symptoms after a road traffic accident. Patients presenting to a hospital emergency department soon after a road traffic accident will be randomly allocated to either the simple cognitive task intervention or usual care. Participants will be followed up at one week and one month. It is predicted that participants given the simple cognitive task intervention will develop fewer flashbacks and less severe clinical symptoms than those who are not. This will inform the potential future development of a simple technique to prevent distressing psychological symptoms after a traumatic event.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over
* Experienced or witnessed a road traffic accident (as a driver, passenger, motorcyclist, cyclist or pedestrian)
* Met the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) criterion A1 for Post-Traumatic Stress Disorder (PTSD) ("experienced, witnessed, or confronted with actual or threatened death or serious injury)
* Can be seen in the emergency department within 6 hours of leaving the scene of the accident
* Report memory of the accident
* Fluent in written and spoken English
* Alert and orientated, Glasgow Coma Scale score (GCS) = 15
* Have sufficient physical mobility to play a computer game on the intervention platform (a Nintendo DS) at the point of taking informed consent
* Willing and able to provide informed consent and complete study procedures
* Willing and able to be contacted following discharge to complete follow-up assessments

Exclusion Criteria:

* Loss of consciousness of > 5 minutes
* Current intoxication
* Report a history of severe mental illness
* Current substance abuse or neurological condition
* Currently suicidal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of flashbacks recorded by participants in a Flashback Record in the week after the accident | Within one week after the accident (Flashback Record will be returned to a researcher at one week follow-up)

SECONDARY OUTCOMES:
Post-traumatic Stress Diagnostic Scale (PDS) | One week and one month follow-up
Impact of Event Scale - Revised (IES-R) | One week and one month follow-up
Hospital Anxiety and Depression Scale (HADS) | One week and one month follow-up

OTHER OUTCOMES:
Feedback Questionnaire | One month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Lalitha Iyadurai, Principal Investigator — University of Oxford; Emily A Holmes, Principal Investigator — MRC Cognition and Brain Sciences Unit, Cambridge
Locations (1):
- Emergency Department, John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom